CLINICAL TRIAL: NCT03823742
Title: Do Biomarkers Predict Response to a Pediatric Chronic Pain Symptom Management Program?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Robert Shulman, M.D., Professor, Baylor College of Medicine
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-43391
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Irritable Bowel Syndrome; Functional Abdominal Pain Syndrome; Functional Gastrointestinal Disorders; Functional Bowel Disorder; Functional Abdominal Pain; Functional Abdominal Pain Disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases | interventions — Cognitive Behavioral Therapy; FODMAP Diet

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized trial with a two group design. Children will be equally likely to be randomized to either CBT or a low FODMAP diet. There is no placebo treatment and no healthy controls are to be studied. Subjects will be stratified based on age (7-9 vs 10-12), sex, baseline pain (mean pain frequency: less than or equal to 50% of the rated intervals or > 50% of the rated intervals, as reported on the baseline pain and stool diary) and PedsQL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy
  Interventions: Other: Cognitive Behavioral Therapy
- Low FODMAP diet (Experimental): Low FODMAP diet
  Interventions: Other: Low FODMAP Diet

INTERVENTIONS:
Other: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT): Study treatments for the child will be conducted by a psychologist or master's level therapist. Therapists will be provided with a standardized protocol for each session . CBT treatment will be given over 1 hour, once a week, for three weeks .
  Arms: Cognitive Behavioral Therapy
Other: Low FODMAP Diet — Low FODMAP Diet Condition: Subjects will receive detailed education by a dietitian about following a low FODMAP diet including a definition of FODMAPs, how to select low FODMAP foods, and how to read food labels to identify FODMAPS. The dietitian will contact the family for 1 hour, once a week, for three weeks.
  Arms: Low FODMAP diet

SUMMARY:
The purpose of this study is find out if we can use simple tests (biomarkers) to tell us if a specific child would benefit most from CBT or from the low FODMAPs diet.

DETAILED DESCRIPTION:
AIM 1: We will categorize children ages 7-12 yrs. of age with FGIDs (n=250) as to whether they have/do not have one or more of the following abnormal physiologic changes: a) Autonomic Nervous System imbalance as indicated by low heart rate variability; and/or (b) Abnormalities in gut physiology: Impaired gut barrier function (increased permeability); and/or increased abundance of species of Gammaproteobacteria and/or Clostridia; and/or Gut neuroimmune dysfunction (increased fecal chromogranin A and secretogranin 2 concentrations).

AIM 2: Children will be randomized to the two treatments most commonly used in clinical practice: CBT or a low FODMAP diet for a 3-week treatment period. We will compare the response to the treatments in those with/without abnormal physiologic biomarkers at 3 weeks, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* A child 7-12 years of age with a FGID will be recruited if the medical evaluation reveals no organic reason for the abdominal pain and the child has abdominal pain that meets the definition of a FGID (i.e., IBS, functional abdominal pain) according to the pediatric Rome III criteria (Rome IV will be substituted when validated). Parents and children must speak and understand English because of the psychological assessment and CBT requirements.

Exclusion Criteria:

* Children who have: had past bowel surgery; documented GI disorders (e.g., Crohn's disease); a serious chronic medical condition (e.g., diabetes); weight and/or height < 2 SD for age; chronic conditions with GI symptoms (e.g., cystic fibrosis); autism spectrum disorder, significant developmental delay, psychosis, or a history of bipolar disorder; been treated with antibiotics/probiotics within 2 mo. (because of effects on gut microbiome analysis), and children who for some reason could not be randomized to the low FODMAP diet.Vegetarian; children who are currently on the FODMAP Diet or receiving CBT Children who speak only Spanish are not eligible because the Rome questionnaire and psychological testing are not available in Spanish. Despite this, a large proportion of the children enrolled will be Hispanic.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom Improvement | 3 to 4 weeks
  Abdominal pain frequency or severity

SECONDARY OUTCOMES:
Improvement in quality of life | 3 months
  PedsQL or Functional Disability
Symptom Improvement | 3 months
  Abdominal pain frequency or severity
Improvement in quality of life | 6 months
  PedsQL or Functional Disability
Symptom Improvement | 6 months
  Abdominal pain frequency or severity

OTHER OUTCOMES:
Improvement in quality of life | 3 to 4 weeks
  PedsQL or Functional Disability

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Shulman, MD, Principal Investigator — Baylor College of Medicine; Rona Levy, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Children's Nutrition Research Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No